CLINICAL TRIAL: NCT05142995
Title: Sleep Related Breathing Disorders, Anxiety, Depression and Quality of Life Assessment in Behcet's Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Lecturer of Chest diseases and tuberculosis, Assiut University
Other Study IDs: WGEK1
Record Dates: First submitted 2021-11-20; First posted 2021-12-03 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Behcet Syndrome
Keywords: Behcet Syndrome; Sleep disorders; Anxiety; Quality of life
MeSH Terms: conditions — Behcet Syndrome; Sleep Wake Disorders; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Behcet disease: Hamilton Anxiety Rating Scale Hamilton Depression Rating Scale SF36 questionnaire Epworth sleepiness scale Pittsburgh sleep quality index
- control: Hamilton Anxiety Rating Scale Hamilton Depression Rating Scale SF36 questionnaire Epworth sleepiness scale Pittsburgh sleep quality index

SUMMARY:
Assessment of Sleep-related breathing disorders, anxiety, depression and quality of life in Behcet's disease.

DETAILED DESCRIPTION:
Behçet's disease (BD) was first described by Turkish dermatologist Hulusi Behçet in 1937 as a triad of recurrent oral aphthae, genital ulcerations and relapsing uveitis. Behçet disease (BD) is an inflammatory vasculopathy with multisystemic involvement. The clinical course usually follows a relapsing-remitting course with heterogeneous clinical manifestations.

The complexity of signs and symptoms in BD can disturb an individual's lifestyle by causing limitation in activity. As a result, numerous psychological problems may arise. Furthermore, it was shown in some studies that in patients with BD with fatigue, there was a significant association with impaired quality of life.

Some studies reported the sleep quality in Behcet disease is very poor, and restless legs syndrome, fatigue, depression, anxiety, and activity of Behcet disease could affect to the quality of life.

However, to date, there have been limited studies regarding sleep quality, quality of life, and depression in Behcet disease patients. Extrapolating that Behcet disease, a kind of Vasculitis, also affects the sleep quality, it is considered a meaningful study to compare and analyze the relationship between disease activity and sleep quality, quality of life, and depression in Egyptian population of Behcet disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical examination and assessment of Behçet's disease activity (International Criteria for Behçet's disease - point score system: scoring ⩾4 indicates Behçet's disease).

Exclusion Criteria:

* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Behçet's disease (BD) patients presented with a triad of recurrent oral aphthae, genital ulcerations and relapsing uveitis. Behçet disease (BD) is an inflammatory vasculopathy with multisystemic involvement. The clinical course usually follows a relapsing-remitting course with heterogeneous clinical manifestations. diagnosis made by International Criteria for Behçet's disease - point score system: scoring ⩾4 indicates Behçet's disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
prevalence and type of sleeping disorders among Behcet's disease population | 4 months
  Pittsburgh Sleep Quality Index (PSQI):
  Self-reported questionnaire consists of a combination of Likert-type and open-ended questions. Scores for each question range from 0 to 3. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, with higher scores indicating more acute sleep disturbances.
presence and degree of anxiety in those patients | 4 months
  Hamilton Anxiety Rating Scale (HAM-A):
  consists of 14 items, each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where a score ≤ 17 indicates mild anxiety, 18-24 mild to moderate severity, and more than 24 moderate to severe anxiety.
presence and degree of depression in those patients | 4 months
  Hamilton Depression Rating Scale (HAM-D):
  The original HAM-D has 21 items, but scoring is based only on the first 17. Scores less than or equal to 7 indicates normal response, 8-13 mild depression, 14-18 Moderate, 19-22 severe, and more than 22 very severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Gamal elddin, Phd, Principal Investigator — Assiut university hospitals
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yazici H, Seyahi E, Hatemi G, Yazici Y. Behcet syndrome: a contemporary view. Nat Rev Rheumatol. 2018 Jan 24;14(2):119. doi: 10.1038/nrrheum.2018.3. PMID 29362466
- [Background] Uygunoglu U, Benbir G, Saip S, Kaynak H, Siva A. A polysomnographic and clinical study of sleep disorders in patients with Behcet and neuro-Behcet syndrome. Eur Neurol. 2014;71(3-4):115-9. doi: 10.1159/000355277. Epub 2014 Jan 21. PMID 24457203
- [Background] International Team for the Revision of the International Criteria for Behcet's Disease (ITR-ICBD). The International Criteria for Behcet's Disease (ICBD): a collaborative study of 27 countries on the sensitivity and specificity of the new criteria. J Eur Acad Dermatol Venereol. 2014 Mar;28(3):338-47. doi: 10.1111/jdv.12107. Epub 2013 Feb 26. PMID 23441863